CLINICAL TRIAL: NCT02173717
Title: Relative Bioavailability of Single Doses of 150 mg Dabigatran Etexilate (Capsule)When Administered Alone, After Seven Days of Dosing With 600 mg Rifampicin(Tablet), and Seven Days and Fourteen Days After Last Administration of Rifampicin in Healthy Male and Female Volunteers (an Open Label, Fixed Sequence, Phase I Study)
Brief Title: Relative Bioavailability of Single Doses of Dabigatran Etexilate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.100
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Rifampin

ARMS (1):
- Dabigatran etexilate (Experimental): Four treatments of 150 mg Dabigatran etexilate (single oral administration) in a fixed sequence.
  1. Single oral administration of dabigatran etexilate on Day 1;
  2. Oral administration of 600 mg rifampicin q.d. in the evening for 7 days (Days 2 to 8) followed by an oral morning dose of dabigatran etexilate on Day 9;
  3. Single oral administration of dabigatran etexilate on Day 16, after 7 days of rifampicin washout;
  4. Single oral administration of dabigatran etexilate on Day 23, after 14 days of rifampicin washout
  Interventions: Drug: Dabigatran etexilate; Drug: Rifampicin

INTERVENTIONS:
Drug: Dabigatran etexilate — 150 mg Dabigatran etexilate
  Other Names: Pradaxa®; BIBR 1048 MS
Drug: Rifampicin — 600 mg Rifampicin
  Other Names: Rifa® 600

SUMMARY:
Study to investigate whether and to what extent the suggested P-glycoprotein (P-gp) inducer rifampicin affects plasma exposure of dabigatran.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the following criteria: based upon a complete medical history, including the physical examination, vital signs (BP, pulse rate), 12-lead ECG, clinical laboratory tests
* Age ≥18 and Age ≤45 years
* Body Mass Index (BMI) ≥18.5 and ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

* Any gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Subjects who in the investigator's judgement were perceived as having an increased risk of bleeding, for example because of:

  * Hemorrhagic disorders or bleeding diathesis
  * Occult blood in faeces or haematocryal
  * Trauma or surgery within the last month or as long as an excessive risk of bleeding persisted after these events, or planned surgery during trial participation
  * History of arteriovenous malformation or aneurysm
  * History of gastroduodenal ulcer disease, gastrointestinal haemorrhage, and haemorrhoids
  * History of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intraarticular bleeding
  * Use of drugs that may have interfered with haemostasis during trial conduct (e.g. acetylic salicylic acid or other non-steroidal anti-inflammatory drugs)
  * Relevant surgery of gastrointestinal tract
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator
* Use of drugs which might have reasonably influenced the results of the trial based on the knowledge at the time of protocol preparation within four weeks prior to administration or during the trial, especially inhibitors or inducers of P-gp, CYP3A4, CYP2C9, or CYP2C19 trial (comment: CYP3A4 inhibitors are for example azole antimycotics, macrolides or grapefruit juice, CYP3A inducers are for example St. John's Wort or certain anticonvulsants)
* Intake of medication, which influences the blood clotting, i.e. acetylsalicylic acid, nonsteroidal anti-rheumatic drugs, cumarin, etc. within 14 days prior to screening or during the trial
* Participation in another trial with an investigational drug within one month prior to administration or during the trial
* Alcohol abuse (more than 60 g/day in males, more than 40 g/day in females)
* Drug abuse
* Blood donation (more than 100 mL within 4 weeks prior to administration)
* Any laboratory value outside the reference range that was of clinical relevance
* Inability to comply with dietary regimen of study centre
* Previous intake of rifampicin
* For female subjects:

  * Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
  * No adequate contraception in women of childbearing potential
  * Lactation period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve over the time interval from 0 extrapolated to infinity (AUC0-inf) of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Maximum measured concentration (Cmax) of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 334hours after treatment on Day1, 9, 16 and 23

SECONDARY OUTCOMES:
AUC0-inf of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Cmax of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Cmax of dabigatran etexilate | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Time from dosing to the maximum concentration (tmax) of dabigatran etexilate | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Cmax of BIBR 1087SE | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
tmax of BIBR 1087SE | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Cmax of BIBR 951BS | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
tmax of BIBR 951BS | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Area under the concentration-time curve over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
AUC0-tz of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Area under the concentration-time curve over the time interval from timepoints t1 to t2 (AUCt1-t2) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
AUCt1-t2 of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Area under the concentration-time curve over the time interval from 0 to 24 h (AUC0-24) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
AUC0-24 of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
tmax of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
tmax of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Terminal rate constant (λz) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
λz of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Terminal half-life (t1/2) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
t1/2 of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Mean residence time after oral administration (MRTpo) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
MRTpo of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Apparent clearance after extravascular administration (CL/F) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
CL/F of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) of free dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Vz/F of total dabigatran | 30 min pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 34 hours after treatment on Day1, 9, 16 and 23
Amount that is eliminated in urine from the time interval 0- 24h (Ae0-24) of total dabigatran | Day 1 and 9
Fraction excreted unchanged in urine from time point 0-24h (fe0-24) of total dabigatran | Day 1 and 9
Renal clearance from the time point 0 until the point 0-24h (CLR, 0-24) of total dabigatran | Day 1 and 9
Ratio of 6-ß-hydroxycortisol/cortisol in morning spot urine as a marker of CYP 3A induction | Day 1 and 9